CLINICAL TRIAL: NCT00547924
Title: Transoesophageal Echocardiography in Liver Transplantation: Left Ventricular Function During Reperfusion
Brief Title: Transoesophageal Echocardiography in Liver Transplantation
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: StV 11-2006
Record Dates: First submitted 2007-10-22; First posted 2007-10-23 (Estimated); Last update posted 2014-04-10 (Estimated); Status verified 2014-04

CONDITIONS: End Stage Liver Disease
MeSH Terms: conditions — End Stage Liver Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Transoesophageal echocardiography — Transoesophageal echocardiography in liver transplantation: left ventricular function during reperfusion

SUMMARY:
Severe hypotension during reperfusion in liver transplantation is a frequent adverse event. Rare data exist so far about pathophysiology of this phenomenon. The exact role of left ventricular function, which might be impaired causing hypotension, has not been elucidated during the period of reperfusion.

Goal of this study is to:

* perform transesophageal echocardiography in order to assess systolic and diastolic left ventricular function during reperfusion
* determine inflammatory mediators in the plasma which could cause left ventricular dysfunction

ELIGIBILITY:
Inclusion criteria:

* Patients on waiting list for liver transplantation.
* Age: 18-75 years.

Exclusion criteria:

* Strictures, tumours and diverticula of the oesophagus.
* History of oesophageal varices with recent bleeding.
* Oesophageal varices and prothrombin time less than 20% or platetlets les than 30000/ml.
* Instable cervical spine.
* Involvement in other studies.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients on waiting list for liver transplantation
Sampling Method: Probability Sample
Enrollment: 17 (Estimated)
Dates: Start 2006-04; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marco Zalunardo, MD, Principal Investigator — UniversitaetsSpital Zuerich
Locations (1):
- University Hospital Zurich, Institute for Anesthesiology, Zurich, Switzerland

REFERENCES:
- [Derived] Zalunardo MP, Schlapfer M, Beck-Schimmer B, Seifert B, Spahn DR, Bettex D. Impact of cytokine release on ventricular function after hepatic reperfusion: a prospective observational echocardiographic study with tissue Doppler imaging. BMC Anesthesiol. 2015 Jul 25;15:107. doi: 10.1186/s12871-015-0080-2. PMID 26209332